CLINICAL TRIAL: NCT03869398
Title: Does Preoperative Calcium and Calcitriol Decrease Rates of Post Thyroidectomy Hypocalcemia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-048
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Hypocalcemia; Thyroid Diseases
MeSH Terms: conditions — Hypocalcemia; Thyroid Diseases | interventions — Calcium Carbonate; Calcitriol

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in the study during their pre-operative consultation with the surgeon once they have been cleared to undergo total thyroidectomy per the usual screening process. The attending surgeon or an IRB approved co investigator will perform the informed consent process (see designated co-investigators). This process will occur in the General Surgery clinic when potential subjects have their 30 minute scheduled preoperative appointment prior to going to the operating room. This process will be conducted in the same manner as the informed consent process for the operation. The nature of their condition will be discussed; the potential risks and benefits of the study will be explained to subjects. The options including not enrolling, enrolling now, and the option to withdraw from the study at any time for any reason will be explained to subjects as well. Once they have consented a consent form will be signed and the subject provided a copy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm: No pre-op medications (No Intervention): patients undergoing total thyroidectomy are started on calcitriol 0.25mcg PO BID and Tums 1,500mg PO TID immediately postoperatively. No pre-operative medications are given
- Intervention arm: Tums and Calcitriol pre-op (Experimental): patients start calcitriol 0.25mcg PO BID and Tums 1,500mg PO TID 5 days before surgery. The five days is determined due to the time it takes vitamin D to have an effect on the guts reabsorption of calcium.
  Interventions: Dietary Supplement: Tums; Dietary Supplement: Calcitriol

INTERVENTIONS:
Dietary Supplement: Tums — start their calcitriol 0.25mcg PO BID and Tums 1,500mg PO TID 5 days before surgery. The five days is determined due to the time it takes vitamin D to have an effect on the guts reabsorption of calcium.
  Arms: Intervention arm: Tums and Calcitriol pre-op
Dietary Supplement: Calcitriol — start their calcitriol 0.25mcg PO BID and Tums 1,500mg PO TID 5 days before surgery. The five days is determined due to the time it takes vitamin D to have an effect on the guts reabsorption of calcium.
  Arms: Intervention arm: Tums and Calcitriol pre-op

SUMMARY:
The investigators are performing this study to determine if supplementation with calcium and calcitriol (vitamin D) before surgery decreases the rate of hypocalcemia (low calcium) after surgery.

Postoperative hypocalcemia (low calcium) is the most common complication after thyroidectomy. Symptoms range from numbness/tingling around the mouth and fingers to severe problems such as low blood pressure, irregular heartbeat, muscle cramps and uncontrollable muscle spasms.

The current standard of practice at Lahey for patients undergoing total thyroidectomy is to start Tums 1500mg three times daily and Calcitriol 0.25mcg twice daily immediately after surgery. Also current practice is for each patient to have their calcium and albumin levels checked at 8 hours and 24 hours after surgery. If the corrected calcium level drops below 8.5 or they exhibit symptoms of hypocalcemia the dose of the Tums and Calcitriol are increased per protocol. All patients must also follow up in 3-4 days to have their calcium and albumin levels rechecked.

The investigators propose to change the above standard practice at Lahey by making only one change. The investigators wish to start Tums and Calcitriol 5 days before surgery, as opposed to after surgery. This will be the only change to the current standard of care at Lahey.

The investigators hypothesize that initiating Tums and Calcitriol supplementation in the preoperative period will decrease the overall rate of postoperative hypocalcemia and its related symptoms. This will possibly decrease length of hospital stay, decrease cost, and prevent any serious complications associated with low calcium.

DETAILED DESCRIPTION:
The main objective of this study is to determine if treating patients with calcitriol and calcium prior to thyroidectomy decreases postoperative hypocalcemia. The primary outcome to be measured is clinical hypocalcemia, defined as peri-oral numbness and/or tingling, numbness and/or tingling in fingers, tetany, seizures, hypotension, palpitations. A secondary outcome measure of biochemical hypocalcemia will be measured. Biochemical hypocalcemia will be defined as a corrected calcium for albumin of less than 8.5 at 8 hours, 1 day, and 3 days postoperatively. Additional secondary outcome measures will be hospital length of stay, need for calcium gluconate IV supplementation, need for additional calcium monitoring.

Postoperative hypocalcemia is the most common complication after thyroidectomy. Symptoms range from perioral numbness/tingling and tingling in fingers to severe complications such as hypotension, arrhythmias and tetany. In prior studies hypocalcemia after thyroidectomy can occur up to 50% of the time. A retrospective cohort study from 2017 shows that treating patients with vitamin D and calcium preoperatively decreases the rate of postoperative hypocalcemia. Preoperative treatment in that study included calcitriol 0.25mcg PO BID and Tums 1,500mg PO TID starting 5 days before surgery. This showed a significant decrease in postoperative hypocalcemia, decreased hospital stay, and overall decrease in cost for patients undergoing total thyroidectomy. This study was limited by its retrospective and observational nature. By performing a prospective randomized study on preoperative supplementation the investigators hope to provide a stronger level of evidence to support this practice.

ELIGIBILITY:
Inclusion Criteria:

* All patients, age >18, undergoing total thyroidectomy are eligible.

Exclusion Criteria:

* partial thyroidectomy, lobectomy, or concurrent parathyroidectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical Hypocalcemia | 3 days post operative
  The main objective of this study is to determine if treating patients with calcitriol and calcium prior to thyroidectomy decreases postoperative hypocalcemia. The primary outcome to be measured is clinical hypocalcemia, defined as peri-oral numbness and/or tingling, numbness and/or tingling in fingers, tetany, seizures, hypotension, palpitations

SECONDARY OUTCOMES:
Biochemical hypocalcemia | 3 days post operative
  A secondary outcome measure of biochemical hypocalcemia will be measured. Biochemical hypocalcemia will be defined as a corrected calcium for albumin of less than 8.5 at 8 hours, 1 day, and 3 days postoperatively
Length of stay | 3 days post operative
  hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: David Brams, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be managed by Co-investigators on a secure spread sheet in a password protected folder on the Lahey General Surgery shared drive. Subjects will be assigned a number and there will be no identifying information on this spreadsheet.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Testa A, Fant V, De Rosa A, Fiore GF, Grieco V, Castaldi P, Persiani R, Rausei S, D'ugo D, De Rosa G. Calcitriol plus hydrochlorothiazide prevents transient post-thyroidectomy hypocalcemia. Horm Metab Res. 2006 Dec;38(12):821-6. doi: 10.1055/s-2006-956504. PMID 17163358
- [Background] Roh JL, Park CI. Routine oral calcium and vitamin D supplements for prevention of hypocalcemia after total thyroidectomy. Am J Surg. 2006 Nov;192(5):675-8. doi: 10.1016/j.amjsurg.2006.03.010. PMID 17071205
- [Background] Reeve T, Thompson NW. Complications of thyroid surgery: how to avoid them, how to manage them, and observations on their possible effect on the whole patient. World J Surg. 2000 Aug;24(8):971-5. doi: 10.1007/s002680010160. PMID 10865043
- [Background] Pattou F, Combemale F, Fabre S, Carnaille B, Decoulx M, Wemeau JL, Racadot A, Proye C. Hypocalcemia following thyroid surgery: incidence and prediction of outcome. World J Surg. 1998 Jul;22(7):718-24. doi: 10.1007/s002689900459. PMID 9606288
- [Background] Maxwell AK, Shonka DC Jr, Robinson DJ, Levine PA. Association of Preoperative Calcium and Calcitriol Therapy With Postoperative Hypocalcemia After Total Thyroidectomy. JAMA Otolaryngol Head Neck Surg. 2017 Jul 1;143(7):679-684. doi: 10.1001/jamaoto.2016.4796. PMID 28418509
- [Background] Iglesias P, Diez JJ. Endocrine Complications of Surgical Treatment of Thyroid Cancer: An Update. Exp Clin Endocrinol Diabetes. 2017 Sep;125(8):497-505. doi: 10.1055/s-0043-106441. Epub 2017 Apr 25. PMID 28444664
- [Background] Docimo G, Ruggiero R, Casalino G, Del Genio G, Docimo L, Tolone S. Risk factors for postoperative hypocalcemia. Updates Surg. 2017 Jun;69(2):255-260. doi: 10.1007/s13304-017-0452-x. Epub 2017 Apr 25. PMID 28444542
- [Background] Falk SA, Birken EA, Baran DT. Temporary postthyroidectomy hypocalcemia. Arch Otolaryngol Head Neck Surg. 1988 Feb;114(2):168-74. doi: 10.1001/archotol.1988.01860140066023. PMID 3337775
- [Derived] Donahue C, Pantel HJ, Yarlagadda BB, Brams D. Does Preoperative Calcium and Calcitriol Decrease Rates of Post-Thyroidectomy Hypocalcemia? A Randomized Clinical Trial. J Am Coll Surg. 2021 Jun;232(6):848-854. doi: 10.1016/j.jamcollsurg.2021.01.016. Epub 2021 Feb 23. PMID 33631337